CLINICAL TRIAL: NCT06765915
Title: Avapritinib Maintenance Following Allogeneic Hematopoietic Stem Cell Transplantation in Acute Myeloid Leukemia With KIT Mutations
Brief Title: Avapritinib Maintenance for AML With KIT Mutations
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-BMT-011
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: AML, Adult
Keywords: AML; KIT mutation; avapritinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Allo-HSCT recipients will begin maintenance therapy with oral Avapritinib tablets at a dose of 100 mg/day, starting 2-4 months post-transplantation. Each treatment cycle lasts 28 days, and therapy will continue for up to 2 years or until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib — After allo-HSCT, CBF-AML patients who have kit mutation would receive avapritinib for maintenance therapy.
  Other Names: KIT inhibitor

SUMMARY:
A multicenter, single-arm clinical study of evaluate the efficacy and safety of avapritinib as maintenance therapy following allogeneic hematopoietic stem cell transplantation for acute myeloid leukemia patients with KIT mutation.

DETAILED DESCRIPTION:
It has been reported that in patients with CBF-associated acute myeloid leukemia (CBF-AML), c-kit mutations occur preferentially in patients with core-binding factor ((8; 21) and inv(16) or t(16; 16) (referred to as inv(16)) rearrangements. However, c-KIT gene mutations, which occur more frequently in patients with CBF-AML, have an incidence of 10% to 45%, which in turn leads to relapse, suggesting a poor prognosis. Nearly 50% of AML patients with concomitant t(8;21) have the c-KIT-D816 mutation. Among AML patients with t(8; 21), patients with c-KIT D816 mutation had significantly shorter OS and EFS than those without this mutation.

Avapritinib, is a novel inhibitor of KIT and PDGFRA-activating ring mutants and a potent and selective inhibitor of KIT D816V, and preclinical studies have demonstrated that compared to Midostauin, Avapritinib is 10-fold more potent against this mutant kinase was 10-fold more potent. A retrospective study [ 14 ] analyzed the efficacy of Avapritinib in patients with t (8;21) AML with KIT mutations who failed allo-HSCT treatment. Among the 13 patients in the D816 mutation, 8 cases reduced RUNX1-RUNX1T1 transcript levels by ≥1 log after 1 month of treatment, and 3 cases turned negative. However, whether avapritinib is effective for maintenance therapy in CBF-AML patients who harbor KIT mutations is unknown.

There is a lack of prospective, controlled studies to clarify the efficacy and safety of XPO1 inhibitor combined with venetoclax as maintenance therapy after allo-HSCTin patients with intermediate- to high-risk AML/MDS, especially those with out specific gene mutation which would be targeted with commerically available inhibitors. Therefore, this multicenter, single-arm study is designed to assess the efficacy and safety of avapritinib as maintenance therapy in CBF-AML patients who harbor KIT mutations after allo-HSCT, with the aim of providing a reference for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 14 years old;
* First allo-HSCT for AML (including secondary AML) ;
* KIT mutation at diagnosis (no restriction on locus for kit mutation
* CR and negative MFC-MRD prior to initiation of maintenance therapy;
* Absolute neutrophil count ≥ 1.0 x 109 /L, platelets ≥ 75 x 109 /L, hemoglobin ≥ 80 g/L before maintenance;
* Normal functioning of major organs and laboratory findings in accordance with the following criteria:AST and ALT) ≤ 3x ULN; Total serum bilirubin ≤ 1.5x ULN unless the patient has Gilbert syndrome; patients with Gilbert-Meulengracht syndrome with bilirubin ≤ 3.0 times the upper limit of normal and direct bilirubin ≤ 1.5 times the upper limit of normal may be included; HB ≥ 70 g/L (had not received a red blood cell transfusion within 1 week prior to administration); ANC ≥ 0.8 x 10^9/L (had not received long-acting colony-stimulating factor (LACSF) within 1 week prior to administration and short-acting colony-stimulating factor (SACSF) within 3 days prior to administration); Platelet count ≥ 20 x 10^9/L (had not received a platelet transfusion within 1 week prior to administration); serum creatinine ≤ 1.5x ULN or creatinine clearance ≥ 60 mL/min; Coagulation function: International Normalized Ratio (INR) ≤1.5×ULN, Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN; Left ventricular ejection fraction (LVEF) ≥45%;
* ECOG PS 0-2 points;
* Expected survival ≥ 3 months;
* Patient consent

Exclusion Criteria:

* concurrently receiving other targeted therapies for AML;
* Prior treatment with a TKI inhibitor that proved ineffective;
* with concurrent FLT3-ITD mutations at enrollment;
* Acute/chronic graft-versus-host disease requiring systemic immunosuppressive therapy prior to maintenance therapy;
* Accompanied by other malignant tumors requiring treatment;
* Have important organ-based diseases: e.g., myocardial infarction, chronic cardiac insufficiency, decompensated hepatic insufficiency, renal failure;
* Active, uncontrolled infection;
* HIV-positive, active hepatitis B (HBV) or active hepatitis C (HCV) requiring antiviral therapy;
* Other interventional clinical studies have been enrolled;
* Men and women of childbearing potential are unwilling to use contraception during and for 12 months after treatment;
* The investigator believes that there are other conditions that make the patient unsuitable for participation in this study.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of relapse | through study completion, an average of 2 year
  disease relapse

SECONDARY OUTCOMES:
Overall survival | through study completion, an average of 2 year
  death as a result of any causes
Non relapse mortality | through study completion, an average of 2 year
  death without disease progression or relapse

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided